CLINICAL TRIAL: NCT00777972
Title: A Bioequivalence Study of Test and Reference Fosinopril Sodium/ Hydrochlorothiazide 20/12.5 mg Tablets Under Fasting Conditions
Brief Title: Bioequivalence Study of Fosinopril Sodium/ Hydrochlorothiazide 20/ 12.5 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B035501
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets fasting conditions
MeSH Terms: interventions — Fosinopril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets by Ranbaxy Laboratories Limited
  Interventions: Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets
- 2 (Active Comparator): Monopril ®.-HCT 20-12.5 mg tablets by Bristol-Meyers Squibb following a single oral dose (1 x 20-12.5 mg tablet
  Interventions: Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets

INTERVENTIONS:
Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets

SUMMARY:
The objective of this study was to compare the relative bioavailability of Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets by Ranbaxy Laboratories Limited with that of Monopril ®.-HCT 20-12.5 mg tablets by Bristol-Meyers Squibb following a single oral dose (1 x 20-12.5 mg tablet) in healthy adult subjects under fasting conditions

DETAILED DESCRIPTION:
This study was a single dose, randomized, two period, two treatment, two sequence crossover study design was used to evaluate the relative bioavailability of Fosinopril sodium and hydrochlorothiazide tablet products when dose (1 x 20-12.5 mg) under fasting conditions. The two periods of the study were separated by a washout period of at least a week.

A total of 36 healthy adult subjects were enrolled in the study. Of all the subjects 34 subjects (21 males and 13 females) completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be at least 18 years old
2. Female subjects with negative serum pregnancy test
3. Subject with no clinically significant abnormal lab values at the pre-entry evaluation
4. Subjects with negative or non-reactive urine drug of abuse, hepatitis B, hepatitis C and HIV screening
5. Subject has acceptable ECG
6. Subject has no evidence of underlying disease at the pre-entry physical examination
7. Subject has agreed to undergo at least a 14 day washout period for prescription drugs prior to the first dosing of the study and throughout the periods of blood sample collection
8. Subject has agreed to undergo at least a 7 day washout period for OTC products, herbal medications, etc. prior to the first dosing of the study medication and throughout the periods of blood sample collections
9. Subject agrees to abstain from consuming alcohol for at least 48 hours prior to each dosing and throughout the periods when blood samples are being obtained
10. Subject agrees to abstain from consuming grapefruit, grapefruit juice, or other foods containing grapefruit for at least 48 hours prior to each dosing and throughout the periods when blood samples are being obtained
11. Subject has given a written consent to participate

Exclusion Criteria:

1. Subject has a history of chronic alcohol consumption (during past 2 years) or drug addiction
2. Subject has a history of serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma
3. Subject has a history of allergic responses to the class of drug being tested.
4. Subject has donated any blood and/ or plasma within the last thirty (30) days prior to the first dosing of the study
5. Subject has taken any investigational drug within thirty (30) days prior to the first dosing of the study
6. Female subjects who are pregnant, breast feeding, or likely to be come pregnant during the study. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (eg condom, IUD) of contraception during the course of the study (first dosing until the last blood collection)
7. Female subjects who have used implanted or injected hormonal contraceptives (except Lunelle ® Monthly Injection) anytime during the 6 months prior to study dosing, Lunelle ® Monthly Injection anytime during the 45 days prior to the study dosing, or used oral hormonal contraceptives within 14 days before dosing.
8. Subject with the inability to read and/ or sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-03; Primary Completion 2003-03 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research Inc, Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html